CLINICAL TRIAL: NCT06333509
Title: A Phase 1/2 Open Label Study to Evaluate the Safety and Efficacy of CT071, an Autologous Anti-GPRC5D CAR T, in Relapsed/Refractory Multiple Myeloma (RRMM) or Relapsed/Refractory Primary Plasma Cell Leukemia (RRpPCL)
Brief Title: Anti-GPRC5D CAR-T Cells (CT071) in Participants With RRMM or RRpPCL
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CT071-HM-01
Record Dates: First submitted 2024-02-19; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Multiple Myeloma; Primary Plasma Cell Leukemia
Keywords: CAR-T; Multiple Myeloma; Primary plasma cell myeloma; CT071; GPRC5D; anti-GPRC5D; genetically modified T-cells; hematologic cancer
MeSH Terms: conditions — Multiple Myeloma; Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase 1; Dose escalation followed by dose expansion Phase 2; Single group of each indication will be dosed at the recommended dose level from Phase 1.
Masking Description: N/Ap
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1 (Experimental): Dose Escalation followed a dose expansion.
  Interventions: Biological: CT071
- Phase 2 (Experimental): Single group of patients for each indication (rrMM, RRpPCL).
  Interventions: Biological: CT071

INTERVENTIONS:
Biological: CT071 — a single CAR-T infusion of CT071

SUMMARY:
A Phase 1/2 Open label, multicenter, clinical trial of autologous CAR T-cell therapy targeting GPRC5D, in participants with relapsed/refractory multiple myeloma or relapsed/refractory primary plasma cell leukemia.

DETAILED DESCRIPTION:
This is an open-label, multicenter, Phase 1/2 trial of CT071 in adult participants with relapsed or refractory multiple myeloma (RRMM) or relapsed or refractory primary plasma cell leukemia (RRpPCL).

The study will be conducted in two phases. Phase 1 of the study will be dose escalation followed by dose expansion. After recommended Phase 2 dose is identified in Phase 1, the enrollment of Phase 2 will start. Following consent, enrolled subjects will undergo apheresis to collect cells for manufacture of the CAR-T cells. Following the manufacture of the CAR-T cells, subjects will receive lymphodepletion prior to CAR T-cell infusion. All subjects who complete the study, as well as those who withdraw from the study after receiving CAR T-cell infusion for reasons other than death or meeting the early termination criteria, will be asked to undergo a 15-year long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed consent;
* Age of ≥ 18;
* Willing and able to adhere to trial visit schedule and other protocol requirements
* Received sufficient prior lines of therapy;
* RRMM participants must have received treatment with at least one proteasome inhibitor, one IMiD and CD38 anti body, must be refractory to the last line of therapy, must have achieved a response (PR or better) to a least 1 prior treatment line;
* RRpPCL participants must have received at least one prior line of therapy.
* Participants must have documented diagnosis of RRMM or RRpPCL.
* The participants should have measurable disease.
* Estimated life expectancy > 12 weeks;
* ECOG performance score 0-1;
* Participants should have bone marrow reserve, renal and hepatic functions;
* Sufficient venous access for apheresis collection, and no other contraindications to apheresis;
* Must be able to stop any anticancer therapy for planned apheresis collection
* Women of childbearing age must undergo a serum pregnancy test with negative results before screening, and are willing to use effective and reliable method of contraception for at least 12 months after T cell infusion;
* Men must be willing to use effective and reliable method of contraception for at least 12 months after T cell infusion.

Exclusion Criteria:

* Any significant condition(s), laboratory abnormality or psychiatric illness that would impair the ability of the participant to receive or tolerate the planned treatment or in the opinion of the investigator, participation would not be in the best interest of the participant (eg, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.
* Pregnant or lactating women;
* HIV, active hepatitis C virus (HCV), or active hepatitis B virus (HBV) infection;
* Any uncontrolled active infection;
* AEs from previous treatment that have not recovered;
* Participants who have had anti-GPRC5D targeted agents;
* Participants who have received autologous stem cell transplantation 12 weeks before apheresis;
* Participants who have received allogenic stem cell transplantation within 6 months of apheresis;
* Participants who have graft versus host disease (GvHD);
* Participants who have received steroids within 14 days of apheresis or lymphodepletion;
* Participants who have plasma cell leukemia secondary to multiple myeloma, Waldenström macroglobulinemia, POEMS (polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes) syndrome or clinically significant symptomatic immunoglobulin light chain (AL) amyloidosis with evidence of end-organ damage;
* Participants who have been administered live attenuated vaccine 4 weeks before apheresis or lymphodepletion;
* Participants who are allergic to fludarabine, cyclophosphamide, tocilizumab, dimethyl sulfoxide (DMSO) or CT071;
* Participants who have clinical significant cardiac conditions that researchers believe that participating in this clinical trial may endanger the health of the patients;
* Participants who require supplemental oxygen;
* Participants who have clinically significant pulmonary conditions;
* Participants who are known to have active autoimmune diseases including but not limited to psoriasis, rheumatoid arthritis and other needs of long-term immunosuppressive therapy;
* Participants with malignancies in addition to MM/pPCL;
* Participants who have central nervous system (CNS) metastases or CNS involvement;
* Participants with a history of stroke or seizures within 6 months prior to apheresis;
* Participants who have undergone major surgery 14 days prior to apheresis or within 28 days of CT071 administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Evaluation of the Safety of CT071 and determination of Maximum Tolerated Dose (MTD). | Day 1 - Month 24
  Frequency, type, and severity of AEs (SAEs, AESIs, laboratory abnormalities).
Phase 2: Objective response rate | Day 1 - Month 24
  Objective response rate (ORR) per IMWG by IRC read; percentage of participants achieving confirmed PR or better per IMWG 2016 consensus criteria.

SECONDARY OUTCOMES:
Phase 1 and 2: Evaluate additional clinical efficacy outcomes | Day 1 - Month 24
  Overall Response Rate/Best Overall Response Rate by investigator (by IMWG stringent complete response/sCR, complete response/CR, very good partial response/VGPR, and partial response/PR by IRC and investigator assessment).
Phase 1 and 2: Evaluate additional clinical efficacy outcomes | Day 1 - Month 24
  Duration of Response by IMWG (stringent complete response/sCR, complete response/CR, very good partial response/VGPR, and partial response/PR by IRC and investigator assessment).
Phase 1 and 2: Evaluate additional clinical efficacy outcomes | Day 1 - Month 24
  Progression Free Survival by investigator assessment
Phase 1 and 2: Evaluate additional clinical efficacy outcomes | Day 1 - Month 24
  Overall Survival
Phase 2: Evaluate additional Safety of CT071. | Day 1 - Month 24
  Frequency, type, and severity of AEs (SAEs, AESIs, laboratory abnormalities).
Phase 1 and 2: Assess immunogenicity of CT071 | Day 1 - Month 60
  Percentage of patients with anti-CT071 drug antibodies
Phase 1 and 2: Evaluate PK profile of CT071 | Day 1 - Month 60
  CAR transgene copy peak value
Phase 1 and 2: Evaluate PK profile of CT071 | Day 1 - Month 60
  CAR transgene copy number persistence
Phase 1 and 2: Evaluate PK profile of CT071 | Day 1 - Month 60
  CAR transgene copy AUC